CLINICAL TRIAL: NCT01596075
Title: Safety and Efficacy of Cannabidiol for Grade I/II Acute Graft Versus Host Disease (GVHD) After Allogeneic Stem Cell Transplantation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0388-11-RMC
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Graft Versus Host Disease
Keywords: Cannabidiol; GVHD; Allogeneic transplantation
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral Cannabidiol (Experimental): Patients undergoing allogeneic SCT will receive standard GVHD prophylaxis consisting of a calcineurin inhibitor and methotrexate or mycophenolate mofetil. Patients developing grade I/II acute GVHD will be treated by IV or oral methylprednisolone 1-2 mg/kg/day and oral cannabidiol at a starting dose of 10 mg twice daily. Doses of cannabidiol can be escalated every day according to clinical response to a maximal dose of 600 mg/day,if no significant drug related side effects present (CTCAE3 grade>2). Cannabidiol will be given up to 90 days.
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Cannabidiol will be dissolved in oil to a predefined concentration.Patients developing grade I/II acute GVHD will be treated by IV or oral methylprednisolone 1-2 mg/kg/day and oral cannabidiol at a starting dose of 10 mg twice daily. Doses of cannabidiol can be escalated every day according to clinical response to a maximal dose of 600 mg/day,if no significant drug related side effects present (CTCAE3 grade>2). Cannabidiol will be given up to 90 days.

SUMMARY:
Graft versus host disease (GVHD) is one of the major causes of death in patients undergoing allogeneic hematopoietic stem cell transplantation. Despite prophylactic measures, the incidence of acute GVHD is estimated at 40-60% among patients receiving transplants from HLA-identical sibling donors, and may even reach 75% in patients receiving HLA-matched unrelated transplants. More effective prevention and treatment strategies are needed.

The immunomodulatory and anti-inflammatory properties of Cannabinoids have been shown in animal models of various inflammatory diseases including multiple sclerosis, inflammatory bowel disease and rheumatoid arthritis.

Cannabidiol is a major non-psychoactive cannabinoid, which has potent anti-inflammatory and immunosuppressive effects.

As such, it may be effective for both prevention and treatment of acute GVHD after allogeneic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years
2. Acute GVHD grade I/II
3. No history of psychosis
4. Signed informed concent

Exclusion Criteria:

1. Acute GVHD grade > II
2. History of psychosis
3. History of asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Complete resolution of acute GVHD | within 90 days from start of therapy

SECONDARY OUTCOMES:
Percentage of patients developing chronic GVHD | 12 months
percentage of patients developing > or = grade 3 toxicity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Yeshurun, MD, Principal Investigator — Davidoff cancer center, Beilinson hospital, Rabin Medical Center
Locations (1):
- Davidof Cancer Center, Beilinson hospital, Rabin medical center, Petah Tikva, Israel